CLINICAL TRIAL: NCT03115853
Title: The Effects of Renin Inhibition on Fibrinolytic Balance and Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, James Muldowney, Assistant Director, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 090738
Record Dates: First submitted 2017-03-16; First posted 2017-04-14 (Actual); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCTZ plus Aliskiren then HCTZ and Placebo (Experimental): HCTZ 25 mg plus Aliskiren 150mg for 2weeks. Aliskiren is increased to 300mg for 4 week if 150mg was tolerated.
  Then HCTZ 25 mg po plus Placebo
  Interventions: Drug: Aliskiren 150 mg; Drug: Placebo; Drug: HCTZ; Drug: Aliskiren 300 mg
- HCTZ and Placebo, then HCTZ and Aliskiren (Experimental): HCTZ 25 mg po plus Placebo.
  Then HCTZ 25 mg plus Aliskiren 150mg for 2weeks. Aliskiren is increased to 300mg for 4 week if 150mg was tolerated.
  Interventions: Drug: Aliskiren 150 mg; Drug: Placebo; Drug: HCTZ; Drug: Aliskiren 300 mg

INTERVENTIONS:
Drug: Aliskiren 150 mg — Aliskiren 150 mg daily for 2 weeks
  Other Names: Tekturna
Drug: Placebo — Placebo tablet for Aliskerin
Drug: HCTZ — HCTZ 25mg every day for 18 weeks
Drug: Aliskiren 300 mg — Aliskiren 300 mg for 4 weeks

SUMMARY:
Aliskiren (also called TekturnaTM) is a new drug for high blood pressure. Aliskiren works by blocking the actions of a substance called renin. Renin is a natural substance in the body that raises blood pressure. Renin is believed to contribute to the production of blood clots by increasing the amount of a substance known as Plasminogen Activator Inhibitor or PAI-1. This study will measure how aliskiren changes the amount of PAI-1 in the blood depending on the time of dosing. The purpose of this study is to find out if it is better to take aliskiren in the morning or at night.

DETAILED DESCRIPTION:
Qualifying subjects will be withdrawn from RAAS blockers in a stepwise fashion over one to two weeks. All other blood pressure medications will be continued. If the subject's blood pressure rises above SBP > 170 or DBP > 120 at any time during the study, they will be excluded and the subject will restart their home medication(s).

Week Two - Visit 2 - Post-taper visit: will be issued hydrochlorothiazide (25mg po, qd x 18 weeks, open label). All study medications will be taken daily between 7 and 10 AM. PAI-1 blood sample will be drawn. Pre-menopausal women will schedule this visit for when they have began their cycle.

Week Four- Visit 3 - If their BP (> 120/60 mmHg), potassium (≤ 5.5 meq/dl) and renal function permit (Cr ≤ 1.5 mg/dl), they will be randomized to aliskiren (150 mg po, qd x 2 weeks) or placebo. If applicable, a urine pregnancy test will be done for child bearing age females.

Week Six - Visit 4 - Titration visit: Subjects will return to the GCRC for an interval history, pill count, blood pressure check, and basic metabolic panel. If their BP, potassium and renal function permit, the medication will be increased to aliskiren (300 mg po, qd x 4 weeks) or placebo (double dose). If applicable, a urine pregnancy test will be done for child bearing age females.

Week Eight - Visit 5 - Post-Titration visit: Subjects will return to the GCRC for an interval history, pill count, blood pressure check and basic metabolic panel. If their BP, potassium and renal function permit, they will remain on the current dose of aliskiren.

Week 10 - Visit 6 - Study Day 1 - Patients will be admitted to the GCRC as an inpatient. They will be asked to lie supine for 24 hours with the head of their bed no higher than 10 degrees. They will have an interval history and physical. An IV catheter will be placed. After an initial void, they will begin a 24 hour urine creatinine, sodium and aldosterone. They will have a baseline BMP, high sensitivity C-Reactive Protein (hsCRP) and CBC. They will have blood drawn every 3 hours for PAI-1 antigen levels, plasma renin activity, plasma ACE activity, plasma aldosterone levels, plasma cortisol and melatonin. White blood cells will be harvested in PaxGene tubes for future extraction of white blood cell mRNA. They will be on a eucaloric, low sodium diet. At the end of the study day they will remain on their home medications, HCTZ (25mg po, qd), however they will stop their current blinded study medication (aliskiren or placebo). Subjects will have DNA banked from unused blood buffy coats. If applicable, UA pregnancy test will be performed by CRC nurses on admission.

Washout Period - The reason for the washout period is four-fold. The washout period insures that drug is completely washed out of the system before initiation of placebo in the arm that received aliskiren first. This will allow the study to observe a placebo effect on blood pressure in the "aliskiren first" arm, in the event that there is one. It would also insure that that sufficient time has passed between SD1 and SD 2 to see the effect of placebo on hsCRP in the "aliskerin first" arm. From a safety standpoint, it insures that subjects have more than 8 weeks to recover their blood counts between study days, as a significant amount of blood is drawn on each study day. Fourth, as there is a menstrual variation in Pai-1 levels, it insures that pre-menopausal women participating in the study will be the same phase of their cycle on SD1 and SD2.

Week 12 - Visit 7 - Mid-Washout visit: Subjects will return to the GCRC for an interval history, pill count, blood pressure check. If their BP permits (<170/120 mmHg) they will remain off study medication. If they are anemic (Hgb < 11) they will be started on iron supplementation.

Week 16 - Visit 8 - Post-Washout visit: Subjects will return to the GCRC for an interval history, pill count, blood pressure check, BMP and CBC, if indicated. If BP and renal function permit, the patient will receive their crossover medication (placebo x 2 weeks or aliskiren 150mg po, qd x 2 weeks). If applicable, a urine pregnancy test will be done for child bearing age females.

Week 18 - Visit 9 - Titration visit 2: Subjects will return to the GCRC for an interval history, pill count, blood pressure check, and basic metabolic panel, and CBC if indicated. If their BP, potassium and renal function permit, the medication will be increased to aliskiren (300 mg po, qd x 4 weeks) or placebo (double dose).

Week 20 - Visit 10 - Post-Titration visit 2: Subjects will return to the GCRC for an interval history, pill count, blood pressure check and basic metabolic pane, and CBC if indicated. If their BP, potassium and renal function permit, they will remain on the current dose of aliskiren. If their Hgb ≥ 11 mg/dl, they will be able to participate in the final study day.

Week 22 - Visit 11 - Study Day 2: Patients will be admitted to the GCRC as an inpatient. They will be asked to lie supine for 24 hours with the head of their bed no higher than 10 degrees. They will have an interval history and physical. An IV catheter will be placed. After an initial void, they will begin a 24 hour urine creatinine, sodium and aldosterone. They will have a baseline BMP, hsCRP, and CBC. They will have blood drawn every 3 hours for PAI-1 antigen levels, plasma renin activity, plasma ACE activity, plasma aldosterone levels, plasma cortisol and melatonin. White blood cells will be harvested in PaxGene tubes for future extraction of white blood cell mRNA. They will be on a eucaloric, low sodium diet. At the end of the study day they will remain on their home medications, and resume home medications that were previously stopped for study purposes. If applicable, UA pregnancy test will be performed by CRC nurses on admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 with hypertension

  * Hypertension is defined as a systolic blood pressure at screening of ≥ 140, a diastolic blood pressure of ≥ 90, or a preexisting diagnosis of hypertension taking antihypertensive medication. If the subject is on anti-hypertensive medication, they can be included in the study, independent of the screening blood pressure.

Exclusion Criteria:

* Serum potassium > 5.0 mmol/L (at the visit directly preceding Randomization)
* History of any cardiovascular event (stroke, TIA, MI, unstable angina, CABG, percutaneous coronary intervention, hospitalization due to HF) during the 3 months prior to Visit 1 or subsequent to enrollment.
* Malignant Hypertension (at Randomization): any patient with SBP > 170 mmHg or DBP > 120 mmHg
* Congestive heart failure NYHA class III and IV
* Unstable serum creatinine
* Second (II) or third (III) degree heart block without a pacemaker.
* Concurrent potentially life threatening arrhythmia or other uncontrolled arrhythmia.
* Clinically significant valvular heart disease.
* Known renal artery stenosis.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study drugs including, but not limited to, any of the following:
* History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection (patients with previous bariatric surgery > 6 months prior to Visit 1 are allowed to participate).
* Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase.
* Evidence of hepatic disease as determined by any one of the following: SGPT value exceeding 3 x Upper Limit of Normal (ULN) at Visit 1, a history of hepatic encephalopathy, a history of cirrhosis, esophageal varices, or a history of portocaval shunt.
* History of malignancy other than basal cell skin cancer within the past five years.
* Any concurrent life threatening condition with a life expectancy less than 2 years.
* History or evidence of drug or alcohol abuse within the last 12 months.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* History of hypersensitivity to any of the study drugs or to medications belonging to the same therapeutic class as the study drugs as well as known or suspected contraindications to the study drugs.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety.
* Persons directly involved in the execution of this protocol.
* Pregnant or nursing (lactating) women
* Transmeridian travel in the past 6 months
* Screening physical and lab findings consistent with the AHA/ADA metabolic syndrome criteria (3 of the following: BP ≥ 130/85 or on antihypertensive medications, waist size > 40" (m) > 35" (f), Fasting Glucose ≥ 100 mg/dl, Triglycerides ≥ 150 mg/dl, HDL <40 mg/dl (m) <50 mg/dl (f))
* Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VUMC, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data for this study was lost. The total number of participants enrolled/completed was pulled from IRB records. Participant age was between 18-65 per protocol. All participants were enrolled in the United States. No other data is available.
Groups:
- All Participants: all participants enrolled in the study
Period: Overall Study
Arm/Group | All Participants
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data lost
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Difference in Peak Plasma PAI-1 Level
Time Frame: baseline to 18 weeks
Population: data was lost and results are unknown
Groups:
- HCTZ Plus Aliskiren 150mg; HCTZ Plus Aliskiren 300mg: HCTZ 25 mg plus Aliskiren 150mg for 2weeks. Aliskiren is increased to 300mg for 4 week if 150mg was tolerated.
- HCTZ and Placebo: HCTZ 25 mg po plus Placebo.
Arm/Group | HCTZ Plus Aliskiren 150mg | HCTZ Plus Aliskiren 300mg | HCTZ and Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Difference in Mean Plasma PAI-1 Level
Time Frame: baseline to 18 weeks
Population: data was lost and results are unknown
Arm/Group | HCTZ Plus Aliskiren 150mg | HCTZ Plus Aliskiren 300mg | HCTZ and Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Difference in Mean Plasma Aldosterone Levels
Time Frame: baseline to 18 weeks
Arm/Group | HCTZ Plus Aliskiren 150mg | HCTZ Plus Aliskiren 300mg | HCTZ and Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Difference in Mean Changes in Plasma Renin Activity.
Time Frame: baseline to 18 weeks
Arm/Group | HCTZ Plus Aliskiren 150mg | HCTZ Plus Aliskiren 300mg | HCTZ and Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Difference in Mean Plasma Peak Aldosterone Levels
Time Frame: baseline to 18 weeks
Population: data was lost and results are unknown
Arm/Group | HCTZ Plus Aliskiren 150mg | HCTZ Plus Aliskiren 300mg | HCTZ and Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: data was lost; unable to provide information on adverse events
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes